CLINICAL TRIAL: NCT03100994
Title: Post-operative Analgesia Efficacy Using Ultrasound-guided Transmuscular Quadratus Lumborum Block Versus Ultrasound-guided Quadratus Lumborum Type II Block.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wu Hsuan-Cheng, Principal Investigator, Department of Anesthesiology,Tri-ServiceGeneralHospital, Tri-Service General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-105-05-157
Record Dates: First submitted 2017-03-24; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Nerve Block
MeSH Terms: interventions — Bupivacaine; Ultrasonography

STUDY DESIGN:
Intervention Model Description: 3 group: Group A: without intervention; Group B: Ultrasound-guided transmuscular quadratus lumborum block; Group C: Ultrasound-guided quadratus lumborum type II block
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group A (No Intervention): without nerve block
- Group B (Active Comparator): Ultrasound guided transmuscular quadratus lumborum block with 0.125% bupivacaine 30ml
  Interventions: Drug: Bupivacaine; Device: Ultrasound
- Group C (Active Comparator): Ultrasound guided quadratus lumborum type 2 block with 0.125% bupivacaine 30ml
  Interventions: Drug: Bupivacaine; Device: Ultrasound

INTERVENTIONS:
Drug: Bupivacaine — injecting anesthetics to different local
  Other Names: Marcaine
  Arms: Group B; Group C
Device: Ultrasound — Ultrasound guided nerve block
  Other Names: Philp
  Arms: Group B; Group C

SUMMARY:
Post-operative analgesia efficacy using ultrasound-guided transmuscular quadratus lumborum block versus ultrasound-guided quadratus lumborum type II block

DETAILED DESCRIPTION:
The Quadratus Lumborum (QL) Block is an ultrasound-guided technique described by Rafael Blanco in 2007. The nerves to the lower abdominal wall can be anesthetized by injecting local anesthetics between the quadratus lumborum muscle and latissimus dorsi muscle, which is called quadratus lumborum type II block. 〝 Transmuscular quadratus lumborum block demonstrates that injectate spreads over the posterior abdominal wall to the psoas major muscle and includes the upper branches of the lumbar plexus.〞described by Adhikary in 2016. However there are no published reports comparing the 2 techniques. In our study, compared of ultrasound-guided QL2-blocks with transmuscular quadratus lumborum block to investigate analgesic consumption, pain level, opioid related side effects and mobilization.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification (ASA) 1~3
* adequate communication skills
* Body mass index < 32

Exclusion Criteria:

chronic pain neurological illness/ neuropathy contraindication against local anesthetics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 48 hours
  morphine consumption

SECONDARY OUTCOMES:
Severity of postoperative pain via visual analogue pain scale (VAS) | 48 hours
  Total cumulative morphine dose in mg used in the first 48 hours after surgery
Nausea or vomiting | 48 hours
  Severity of nausea or vomiting in the first 48 hours after surgery. Severe :3 Moderate:2 Mild:1 None: 0
time to mobilization | 48 hours
  Time to mobile in the first 48 hours after surgery
Skin itch | 48 hours
  Severity of skin itch in the first 48 hours after surgery. Severe :3 Moderate:2 Mild:1 None: 0

CONTACTS AND LOCATIONS:
Overall Officials: Hsuan-Cheng Wu, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adhikary SD, El-Boghdadly K, Nasralah Z, Sarwani N, Nixon AM, Chin KJ. A radiologic and anatomic assessment of injectate spread following transmuscular quadratus lumborum block in cadavers. Anaesthesia. 2017 Jan;72(1):73-79. doi: 10.1111/anae.13647. Epub 2016 Oct 12. PMID 27730633
- [Result] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488